CLINICAL TRIAL: NCT05339191
Title: A Brief Compassionate Imagery Intervention for People With an Intellectual Disability: A Case Series in a Clinical Setting
Brief Title: Compassionate Imagery for People With An Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lanarkshire (Other Government)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: L19092
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Participants who are attending the NHS Lanarkshire Community Learning Disability Team and are experiencing mental health difficulties will be recruited. Participants will be asked to attend a two-session workshop through which they will be supported to develop and use their own compassionate image. The research questions will be answered by obtaining descriptive data from data recording sheets completed during the sessions and by interviewing participants about their experiences of the workshop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassionate image workshop (Experimental): Participants attend a workshop through which they will be supported to develop and use their own compassionate image.
  Interventions: Behavioral: Compassionate image workshop

INTERVENTIONS:
Behavioral: Compassionate image workshop — Participants attend a workshop through which they will be supported to develop and use their own compassionate image.

SUMMARY:
The current study aims to explore the adaptation of compassionate imagery for people with an intellectual disability who are experiencing mental health difficulties. It will explore whether participants are able to generate and use their own compassionate image, as well as exploring the participants' views of engaging in the workshop. It is an early exploratory study in what is hoped will be a longer process consisting of future feasibility and piloting work.

Between 6-10 participants who are attending the National Health Service (NHS) NHS Lanarkshire Community Learning Disability Team and are experiencing mental health difficulties will be recruited. Participants will be asked to attend a two-session workshop through which they will be supported to develop and use their own compassionate image. The research questions will be answered by obtaining descriptive data from data recording sheets completed during the sessions and by interviewing participants about their experiences of the workshop.

DETAILED DESCRIPTION:
People with an intellectual disability experience widespread stigma, mistreatment and abuse (Scior and Werner, 2016, Gravell, 2012, Hughes et al., 2012, Jones et al., 2012). These are likely to lead individuals to experience shame and self-criticism, which can contribute to the development of mental health difficulties. Indeed, many people with an intellectual disability do experience mental health difficulties (Buckles et al., 2013).

Compassion-Focused Therapy (CFT) is a psychological therapy which aims to reduce shame and self-criticism by developing a person's ability to feel compassion. It involves enabling individuals to learn to soothe themselves when they feel distressed. Compassionate imagery is one CFT technique used to do this (Gilbert, 2009). This can involve developing a mental image of a compassionate person or animal who is wise, strong, warm and non-judgemental.

The individual is encouraged to explore their experience of imagining this, which may include feeling a sense of safety, warmth and connectedness (Gilbert, 2015).

The current study aims to explore the adaptation of compassionate imagery for people with an intellectual disability who are experiencing mental health difficulties. It will explore whether participants are able to generate and use their own compassionate image, as well as exploring the participants' views of engaging in the workshop. It is an early exploratory study in what is hoped will be a longer process consisting of future feasibility and piloting work.

Between 6-10 participants who are attending the NHS Lanarkshire Community Learning Disability Team and are experiencing mental health difficulties will be recruited. Participants will be asked to attend a two-session workshop through which they will be supported to develop and use their own compassionate image. The research questions will be answered by obtaining descriptive data from data recording sheets completed during the sessions and by interviewing participants about their experiences of the workshop.

ELIGIBILITY:
Inclusion Criteria:

* Open to NHS Lanarkshire's Community Learning Disability Team (CLDT) and will therefore be aged 16 or above
* Experiencing mental health difficulties

Exclusion Criteria:

* Do not have capacity to provide informed consent
* Have insufficient communication skills to engage with the tasks
* Have sensory impairments which are likely to inhibit their ability to engage with the study materials
* Actively suicidal
* Likely to be disruptive or distressed in a group setting
* Known to have previously engaged in a piece of therapeutic work involving the development of a compassionate image

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Compassionate image | 6 months
  Number of participants that are able to generate their own compassionate image

SECONDARY OUTCOMES:
Self-soothing | 6 months
  Number of participants that report using their compassionate image to self-soothe outside of sessions and the number that find this to be helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Holm, Principal Investigator — NHS Lanarkshire
Locations (1):
- Kilsyth Community Centre, Kilsyth, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
None will be shared